CLINICAL TRIAL: NCT00999570
Title: High Volume Specialty Knee Replacement Surgeons Achieve Better Clinical and Quality-of-Life Scores
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Tan Sok Chuen, Singapore General Hospital
Other Study IDs: 2009/626/D
Record Dates: First submitted 2009-10-20; First posted 2009-10-22 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Total Knee Arthroplasty
Keywords: outcome; quality of life; total knee arthroplasty; clinical outcome scores post total knee arthroplasty; quality of life scores post total knee arthroplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients operated by AR trained surgeons: patients who had their total knee replacements performed by surgeons who have completed a fellowship training in adult reconstruction surgery
  Interventions: Other: Specialty training for knee surgeons
- Patients operated by non-AR surgeons: patients who had their total knee replacements performed by orthopaedic surgeons who did not complete an adult reconstruction fellowship training

INTERVENTIONS:
Other: Specialty training for knee surgeons
  Groups: Patients operated by AR trained surgeons

SUMMARY:
To determine whether specialty training or high volume of operative experience is associated with better clinical outcome and quality-of-life scores.

DETAILED DESCRIPTION:
Primary total knee replacements are becoming a commonly performed procedure. Many general orthopaedists can perform large numbers of such surgeries. Thus, we aim to find out if there is value of having surgeons with AR fellowship training to perform primary total knee arthroplasty. This has an implication in the direction of the training of future AR surgeons and in the distribution of operative cases.

ELIGIBILITY:
Inclusion Criteria:

* patients who require total knee arthroplasty seen during the specified period

Exclusion Criteria:

* revision total knee arthroplasty
* unicompartmental or bicompartmental knee arthroplasty

Ages: 37 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients seen at Singapore General Hospital who require total knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 3458 (Actual)
Dates: Start 2004-01; Primary Completion 2007-05 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To determine whether specialty training or high volume of operative experience is associated with better clinical outcome and quality-of-life scores. | 2 years

SECONDARY OUTCOMES:
To determine which other factors are predictors of better outcome score and quality-of-life scores. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sok Chuen Tan, MBBS, MRCS, Principal Investigator — Singapore General Hospital; Seng Jin Yeo, FRCS, FAMS, Study Director — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Katz JN, Mahomed NN, Baron JA, Barrett JA, Fossel AH, Creel AH, Wright J, Wright EA, Losina E. Association of hospital and surgeon procedure volume with patient-centered outcomes of total knee replacement in a population-based cohort of patients age 65 years and older. Arthritis Rheum. 2007 Feb;56(2):568-74. doi: 10.1002/art.22333. PMID 17265491